CLINICAL TRIAL: NCT00388128
Title: Effects of Caffeine in Patients With Intermittent Claudication.
Brief Title: Caffeine and Intermittent Claudication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Herning Hospital (Other); Central Jutland Regional Hospital (Other)
Responsible Party: Regional Hospital Herning, Surgical Research Unit
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-001902-10; 2006/168
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Intermittent Claudication
Keywords: Intermittent Claudication; PAD; Caffeine; Walking capacity; ABI; QoL; Growth factor
MeSH Terms: conditions — Intermittent Claudication | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator)
  Interventions: Drug: Caffeine 6mg/kg

INTERVENTIONS:
Drug: Caffeine 6mg/kg — Capsules of caffeine 6 mg/kg, taken orally at each test. Before and after treadmill testing

SUMMARY:
The purpose of this study is to evaluate the change in Walking capacity after an intake of caffeine. The study design is cross-over and follow-up of 80 patients with leg pain caused by narrowing of their leg arteries, Peripheral Vascular Disease (PAD), stage II. Half of all will be revascularised, follow up will be after 3 months. It is hypothesized that caffeine (6mg/kg) can be a cheap, safe drug before walking exercise. Primary endpoint is maximum walking distance (MWD), treadmill-testing,(constant load, 0%,2m/h). Secondary endpoints are pain free walking distance (PWD), maximum muscle strength, endurance, reaction speed, balance, cognitive function, health related quality of life (SF-36).

DETAILED DESCRIPTION:
PAD has a prevalence of 15-20 % in an elderly (>50) western population. PAD can not be seen in isolation but represents the peripheral manifestation of a generalized artherosclerosis. The co-morbidity with coronary or cerebralartherosclerosis depends on the degree of severity of PAD, the relative risk of a death (predominantly cardiac) is increased by a factor 4. From af medical and a socio-economic point of view there is the need to control the PAD complication rate and related treatment costs as effectively as possible.

The aim of any treatment of intermittent claudication is a clinically relevant improvement in the patient´s mobility and quality of life.

There is agreement, that physical training does improve the collateralisation of vascular lesions, the rheologic properties of blood and lead to a shift from glycolytic to oxidative muscle fibers in the working musculature which increases the capillary density. The effect of physical training is also to modify the patients risk factor profile, even moderate training increase the insulin receptor sensitivity and the fibrinolytic activity and decrease the dLDL/HDL ratio and the diastolic blood pressure in hypertensive patients - and thereby decrease the overall cardiac mortality.

This is a Phase 3, 12-week, double-blind, randomized, placebo-controlled cross-over and a follow-up study with 80 patients with intermittent claudication, half of which will be revascularized.

The objectives of this study are to evaluate the efficacy of caffeine (6mg/kg)and the revascularisation procedure. The primary end-point will be maximal walking distance (MWD) in both groups of patients. Other efficacy measures will include claudication onset time (PWD), changes in Ankle Brachial Index (ABI), Quality of Life (QoL), cognitive function, plasma response of Vascular Endothelian Growth Factor (VEGF, FGF). Safety variables will include routine hematology parameters and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* men and women > 40 years
* history of IC of the lower extremities, Fontaine II
* ankle-brachial index (ABI)> 0.9 (subjects who are referred for a revasularizarition procedure)

Exclusion Criteria:

* dementia
* diabetes
* illness or reason to be unable to participate, f.ex. general weakness, amputation or arthritis
* acute illness, f.ex. inflammation, unstable angina
* other reasons which contraindicate participation/treadmill exercise
* intake of Trental and/or Teofyllamin
* weight > 100kg

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Quality of life | during test 1 and 3
Maximum walking distance | during treadmill test

SECONDARY OUTCOMES:
Painfree Walking Distance | treadmill test
Max muscle strength (MVC) of kneeextension | At end of each test
Endurance of 50%MVC kneeextension | At end of each test
Postural stability | in all tests
Reaction speed | in all tests
Cognitive function | in all tests
Walking Impairment Questionnaire | in first and third test
vascular endothelian growth factors VGF. FGF | before and after 1. and 2. test

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette H Momsen, MPH, Phys, ph.D stud, Principal Investigator — Herning Hospital
Locations (1):
- Herning Hospital, Surgical research dep., Herning, Central Jutland, Denmark

REFERENCES:
- [Derived] Momsen AH, Jensen MB, Norager CB, Madsen MR, Vestersgaard-Andersen T, Lindholt JS. Randomized double-blind placebo-controlled crossover study of caffeine in patients with intermittent claudication. Br J Surg. 2010 Oct;97(10):1503-10. doi: 10.1002/bjs.7149. PMID 20629111